CLINICAL TRIAL: NCT00247052
Title: the Post Operative Pericardial Effusion (POPE) Treatment Study
Brief Title: Non Steroidal Anti Inflammatory Treatment for Post Operative Pericardial Effusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: CLIPA (Unknown); Clinact (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-06
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Pericardial Effusion
Keywords: post operative pericardial effusion; NSAID
MeSH Terms: conditions — Pericardial Effusion | interventions — Diclofenac

ARMS (2):
- diclofenac (Active Comparator): diclofenac
  Interventions: Drug: diclofenac
- 2 (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: diclofenac — diclofenac 50 mg bid versus placebo bid
  Arms: diclofenac
Drug: diclofenac — diclofenac 100 mg per day for 14 days
  Arms: diclofenac
Drug: matching placebo
  Arms: 2

SUMMARY:
The aim of the sudy is to evaluate, through clinical, biological and transthoracic echocardiography follow up, the evolution of post operative (cardiac surgery) pericardial effusion and mostly to evaluate the efficiency of a non steroidal anti inflammatory (NSAID) drug (diclofenac)for this indication.

DETAILED DESCRIPTION:
Following cardiac surgery, the incidence of Pericardial effusion (PE) is high (50-85%) . The risk of tamponade is well acknowledged : about 2%. We published in 2004 in CHEST a study which allows us to know the natural history of post-operative PE and to validate, for the first time the use of an echocardiographic classification for predicting the occurrence of a tamponade. NSAID are widely used in this setting, but no study has ever been conducted trying to assess their efficiency. The aim of the study is therefore obvious : must we use NSAID in order to prevent post operative cardiac tamponades ?.

In order to answer this question, we are going to conduct a double-blind randomized study comparing diclofenac to a placebo.

Every patient hospitalized in a post operative cardiac rehabilitation center less than 30 days after cardiac surgery and presenting at the first TTE (Trans Thoracic cardiac Echography) a PE of severity > 2 (that is to say about 10 % of the totality of the patients having undergone a cardiac operation) will be included.: after randomisation, patients will receive a placebo or diclofenac (50 mg ) bid, in a double blind way, during 14 days.

Trans thoracic cardiac echography, creatininemia, haemoglobinemia, International Normalized Ratio (for patients receiving a vitamin K antagonist) will be performed once a week during 2 weeks.

Clinical assessment will be done every day (there will be no outpatient

Primary end point : evolution of the mean echocardiographic score in each group

-Secondary end-points :

Number of tamponades Number of patients in whom the individual echographic grade is decreasing of at least one point Number of pericardiotomy Creatininemia Haemoglobinemia PE evolution in patients having an inflammatory syndrome (C reactive Protein >30) PE evolution in patients receiving a vitamin K antagonist

86 patients per group are necessary; therefore we will include a total of 200 patients

ELIGIBILITY:
Inclusion Criteria:

* -Every patient hospitalized in a post operative cardiac rehabilitation center less than 30 days after cardiac surgery and presenting at the first TTE (Trans Thoracic cardiac Echography) a PE of severity > or equal to 2 (that is to say loculated effusion >10 millimeters or circumferential effusion > 1 mm ) will be included

Exclusion Criteria:

* Cardiac transplantation
* Age <18 and > 80
* Pregnancy
* Diclofenac contra indication (allergy, gastro intestinal ulcer, renal insufficiency, cardiac failure…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
comparison of the evolution between day 1 and day 14 of the mean echocardiographic score of pericardial effusion between treated and untreated (placebo) groups

SECONDARY OUTCOMES:
Number of tamponades
Number of patients in whom the individual echographic grade is decreasing of at least one point
Number of pericardiotomy
Creatinemia
Haemoglobinemia
PE evolution in patients having an inflammatory syndrome (C reactive Protein >30)
PE evolution in patients receiving a vitamin K antagonist

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Meurin, MD, Principal Investigator — Les grands Prés; 27 rue Sainte Christine 77174 , Villeneuve Saint Denis, France; Philippe Meurin, MD, Principal Investigator — Les Grands Prés
Locations (5):
- France (5):
  - Centre Hospitalier Chateau Lemoine, Bordeaux
  - Hôpital Bligny, Briis-sous-Forges
  - IRIS, Lyon
  - Hôpital Broussais, Paris
  - Les Grands Prés, Villeneuve-Saint-Denis

REFERENCES:
- [Background] Meurin P, Weber H, Renaud N, Larrazet F, Tabet JY, Demolis P, Ben Driss A. Evolution of the postoperative pericardial effusion after day 15: the problem of the late tamponade. Chest. 2004 Jun;125(6):2182-7. doi: 10.1378/chest.125.6.2182. PMID 15189940
- [Derived] Meurin P, Tabet JY, Thabut G, Cristofini P, Farrokhi T, Fischbach M, Pierre B, Driss AB, Renaud N, Iliou MC, Weber H; French Society of Cardiology. Nonsteroidal anti-inflammatory drug treatment for postoperative pericardial effusion: a multicenter randomized, double-blind trial. Ann Intern Med. 2010 Feb 2;152(3):137-43. doi: 10.7326/0003-4819-152-3-201002020-00004. PMID 20124229